CLINICAL TRIAL: NCT04975516
Title: Phase 2 Randomized Trial of Standard of Care Chemotherapy With or Without Stereotactic Body Radiation Therapy for the Treatment of Oligometastatic Pancreatic Adenocarcinoma
Brief Title: Standard of Care Chemotherapy With or Without Stereotactic Body Radiation Therapy for Oligometastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC210711; NCI-2021-07006 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-011610 (Other: Mayo Clinic)
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Stage IV Pancreatic Cancer AJCC v8; Recurrent Pancreatic Adenocarcinoma; Oligometastatic Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy; Radiosurgery; Magnetic Resonance Spectroscopy; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (SBRT, chemotherapy) (Experimental): Patients undergo SBRT QD or every other day for 5 fractions, and receive chemotherapy per standard of care.
  Interventions: Drug: Chemotherapy; Radiation: Stereotactic Body Radiation Therapy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Other: Questionnaire Administration
- Group II (chemotherapy) (Active Comparator): Patients receive chemotherapy per standard of care.
  Interventions: Drug: Chemotherapy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Chemotherapy — Given chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Group I (SBRT, chemotherapy)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized Tomography (CT) scan; CT; CT SCAN
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging (MRI); MRI; Magnetic Resonance / Nuclear Magnetic Resonance; MRI Scan; MRIs; NMRI; nuclear magnetic resonance imaging; sMRI; Structural MRI
Procedure: Biospecimen Collection — Undergo blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the effect of standard of care chemotherapy with or with out stereotactic body radiation therapy in treating patients with pancreatic cancer that has spread to a limited amount of places in the body (oligometastatic). Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Chemotherapy drugs work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy with stereotactic body radiation therapy may help improve tumor control, decrease risk of tumor spreading more, decrease side effects, and prolong survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare progression free survival (PFS) between stereotactic body radiation therapy (SBRT) + standard chemotherapy versus (vs.) standard chemotherapy alone in patients with oligometastatic pancreatic cancer.

SECONDARY OBJECTIVES:

I. Confirmed response rate. II. Overall survival. III. Adverse events. IV. Longitudinal assessment of circulating tumor cells (CTC) and circulating tumor deoxyribonucleic acid (ctDNA).

CORRELATIVE RESEARCH OBJECTIVE:

I. To evaluate fatigue, and other patient-reported outcomes.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients undergo SBRT once daily (QD) or every other day for 5 fractions and receive chemotherapy per standard of care on study. Additionally, patients undergo computed tomography (CT), magnetic resonance imaging (MRI), and blood collection throughout the study.

GROUP II: Patients receive chemotherapy per standard of care on study. Additionally, patients undergo CT, MRI, and blood collection throughout the study. Patients who have local disease progression at known sites and no new sites of progression may crossover to the radiotherapy arm.

After completion of study treatment, patients are followed up at 7 and 14 days, and then every 8-12 weeks for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histologically confirmed adenocarcinoma of pancreatic origin with pathologic material reviewed by the Department of Pathology at Mayo Clinic, if available and applicable
* Image proven oligometastatic pancreatic cancer patients (i.e., synchronous & metachronous)

  * Oligometastatic defined as: =< 5 extracranial metastatic tumors (brain metastasis patients are excluded; indeterminate lung nodules stable on 2 consecutive imaging studies spaced more than 4 weeks apart will not count as sites of oligometastatic disease)
  * All sites must be amenable to SBRT (positive peritoneal washings cytology or Kras cell free (cf)DNA, and positive peritoneal biopsy would be considered ineligible)
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Non-measurable disease

  * NOTE: Tumor lesions in a previously irradiated area are not considered measurable disease; disease that is measurable by physical examination only is not eligible
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Negative pregnancy test done =< 7days prior to registration, for women of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Willing to provide tissue and/or blood samples for correlative research purposes
* Hemoglobin >= 9.0 g/dL (obtained =< 28 days prior to registration)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 28 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 28 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (If known Gilbert's syndrome, then =< 3.0 x ULN) (obtained =< 28 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3 x ULN (=< 5 x ULN for patients with liver involvement) (obtained =< 28 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) =< 1.5 x ULN OR if patient is receiving anticoagulant therapy and INR or aPTT is within target range of therapy (obtained =< 28 days prior to registration)
* Calculated creatinine clearance >= 45 ml/min using the Cockcroft-Gault formula (obtained =< 28 days prior to registration)

Exclusion Criteria:

* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception
* Any of the following prior therapies:

  * Surgery =< 3 weeks prior to registration
  * Prior radiation to an overlapping area
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 1 year prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix
  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2026-07-02 (Estimated); Study Completion 2027-07-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Time from randomization to the first of either disease progression or death from any cause, assessed up to 2 years
  Disease progression will be determined based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria and will be documented at each enrolling site with no central review planned.

SECONDARY OUTCOMES:
Confirmed response rate | Up to 2 years
  A patient will be classified as a confirmed response per the RECIST 1.1 criteria, if they have a partial or complete response for 2 consecutive evaluations at least 4 weeks apart. The proportion of patients with a confirmed response will be calculated and compared between the 2 arms using a Chi-square or Fisher's Exact test.
Overall survival | Time from study entry to death from any cause, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method, where the log-rank test will be used to compare the 2 treatment arms.
Incidence of adverse events | Up to 2 years
  The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events version 5.0. The frequency and percentage of grade 3+ adverse events will be compared between the 2 treatment arms. Comparisons between arms will be made by using either the Chi-square or Fisher's Exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Rutenberg, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Elhariri A, Patel J, Mahadevia H, Modi K, Albelal D, Majeed U, Jones JC, Borad MJ, Tran NH, Rutenberg MS, Babiker H. Stereotactic body radiation therapy in oligometastatic pancreatic cancer: overall survival improvement and SMAD4 as a predictor of progression-free survival. J Gastrointest Oncol. 2025 Aug 30;16(4):1658-1666. doi: 10.21037/jgo-2025-100. Epub 2025 Aug 26. PMID 40950337
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials